CLINICAL TRIAL: NCT01645696
Title: Three-day, In-clinic, Clamp Evaluation of the BD 2nd Generation Continuous Glucose Sensor in Subjects With Type 1 Diabetes
Brief Title: Three-day, In-clinic Evaluation of the BD 2nd Generation Continuous Glucose Sensor Device in Type 1 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Device Feasibility
Other Study IDs: BDT-11-CGM002
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Diabetes
Keywords: Diabetes; Type 1 Diabetes; Continuous glucose monitoring; Blood glucose; Blood glucose sensor; Glucose Binding Protein (GBP)
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BD Continuous Glucose Monitor (CGM) with outer layer (Experimental): A subcutaneous glucose binding protein sensing device to continuously monitor glucose in diabetics.
  Interventions: Device: BD CGM with Outer Layer
- BD CGM without outer layer (Experimental): A continuous glucose binding protein sensing device used to monitor glucose in Diabetics
  Interventions: Device: BD CGM without Outer Layer
- Medtronic iPro 2 Professional CGM (Active Comparator): Commercial glucose oxidase continuous glucose monitor
  Interventions: Device: Medtronic iPro2 Professional CGM

INTERVENTIONS:
Device: BD CGM with Outer Layer — continuous (every 2 minutes) subcutaneous glucose monitoring for 72 hours.
  Arms: BD Continuous Glucose Monitor (CGM) with outer layer
Device: BD CGM without Outer Layer — continuous (every 2 minutes) subcutaneous glucose monitoring over 72 hours.
  Arms: BD CGM without outer layer
Device: Medtronic iPro2 Professional CGM — continuous subcutaneous glucose monitoring for 72 hours
  Arms: Medtronic iPro 2 Professional CGM

SUMMARY:
The purpose of this study is to investigate the accuracy and performance of a new subcutaneous continuous glucose monitor (BD-CGM, Becton Dickinson) in hyperglycemic (high blood sugar) and hypoglycemic (low blood sugar) "clamp" conditions and during meal excursions over the course of 72 hours as compared to a commercially available monitor.

DETAILED DESCRIPTION:
This is a single site, non-randomized study. The study consists of a Screening Visit (Visit 1) during which the subject will be consented and the inclusion exclusion criteria confirmed. An interventional visit (Visit 2)which consists of a 72 hour in-clinic stay and a Follow-up Visit (Visit 3). Subjects eligible for the study will be admitted to the clinic for the Study Visit 2 in the afternoon on the day before the first Clamp is performed. An IV line for blood sampling will be established. One blood sample will be obtained for glucose determination and a second blood sample will be collected for immunoassay development before any sensors are inserted. Two BD-Glucose Binding Protein-Continuous Glucose Monitor Sensors(BD-GBP-CGM), with and without outer layer, and one commercial CGM sensor will be inserted in the subcutaneous tissue in the abdomen shortly thereafter. Blood sampling intervals will be adjusted over the 3 study days as determined by the study event (i.e. clamp period, meal excursion, nighttime). During the hyper- /hypo-glycemic clamps periods on Day 1 and Day 3 blood samples will be taken more frequently, every 5-10 minutes. During the breakfast meal on Day 2 sampling will occur at 10-15 minute intervals for 4 hours to capture the meal excursion. Sampling will be less frequent during the evening meal and at night during sleep hours.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes mellitus for ≥1 year. For an individual to be enrolled at least one criterion from each list must be met.
2. Criteria for documented hyperglycemia (at least 1 must be met):

   1. Fasting glucose ≥ 7 mmol/L [126 mg/dL] - confirmed
   2. Two-hour OGTT (oral glucose tolerance test) glucose ≥ 11.1 mmol/L [200 mg/dL] - confirmed
   3. HbA1c ≥6.5% documented - confirmed
   4. Random glucose ≥ 11.1 mmol/L [200 mg/dL] with symptoms
   5. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes
3. Criteria for requiring insulin at diagnosis (1 must be met):

   1. Participant required insulin at diagnosis and continually thereafter
   2. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
   3. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
4. Signed informed consent
5. Age ≥18 and ≤65 years old
6. Body mass index between 19 and 35 kg/m2, inclusive
7. HbA1c ≤ 10.0%

Exclusion Criteria:

1. Uncontrolled arterial hypertension (diastolic blood pressure > 90 mm Hg and/or systolic blood pressure > 160 mm Hg)
2. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥ three times the upper reference limit
3. Impaired renal function measured as creatinine > 1.2 times above the upper limit of normal
4. Diabetic ketoacidosis in the past 6 months
5. Severe hypoglycemia resulting in a seizure or loss of consciousness in the 6 months prior to enrollment
6. Conditions which may increase the risk of hypoglycemia or conditions of known microvascular (diabetic) complications will be assessed on an individual basis with exclusion based on the discretion of the principal investigator.
7. Current use of medications containing > 4000 mg acetaminophen per day.
8. Current use of MAO (monoamine oxidase) inhibitors.
9. Known allergy to eggs
10. Pregnancy, breast-feeding or intention of becoming pregnant
11. Current or recent alcohol or drug abuse by subject history.
12. Blood donation of more than 473 ml within the last 56 days
13. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
14. Any skin condition that prevents sensor placement on the abdomen (e.g., bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
15. Known allergy to medical adhesives, e.g. Tegaderm
16. Hematocrit < 38% (males) and < 36% (females)
17. Potassium < 3.4 mmol/L
18. Active enrollment in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 72 hours
  Blood glucose will be measured by the BD-Continuous Glucose Monitor, with and without outer layer, the commercially available Medtronic iPro2 and the YSI (Yellow Springs Instrument) Glucose analyzer (control) for 72 hours. Blood glucose will be used to determine performance of the device to include warm up behavior, lag time and accuracy of the blood glucose monitor over 72 hours.
Number of participants with adverse events | up to 89 days or until the subject is discharged
  At each study contact, subjects will be questioned about any adverse events that may have occurred and are potentially related to the device.

SECONDARY OUTCOMES:
Skin Effects-Draize Scoring for Skin Irritation | Up to 36 days
  Local reaction at insertion sites will be scored for redness and swelling at the following timepoints: Visit 2-pre-insertion of devices, immediately post insertion of the devices, each morning of Day 1, 2 and 3, immediately after removal of the devices and at Visit 3.
Skin thickness using ultrasound | Upon removal of the devices
  Skin thickness will be measured at the sensor sites and a control site (on the abdomen) immediately after removal of the device.
Insulin levels | 72 hours
  Blood samples will be taken at pre-determined times following insulin dosings to test for insulin levels:
antibodies against the glucose binding protein | 36 days
  A blood sample will be taken at the beginning of Visit 2 and at Visit 3 to test for antibody production following exposure to the sensor's glucose binding protein.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Endocrinology Centre, Clinical Research Unit
Locations (1):
- >LMC Endocrinology Centre, Clinical Research Unit, Toronto, Ontario, Canada